CLINICAL TRIAL: NCT02081534
Title: A Phase 2b, Randomized, Double Blind, Placebo-controlled, Parallel Group, Multicentre Dose Finding Study to Evaluate the Efficacy, Safety and Tolerability of AZD1722 to Treat Hyperphosphatemia in End-Stage Renal Disease Patients on Hemodialysis (ESRD-HD)
Brief Title: Dose Finding Study to Treat High Phosphate Levels in the Blood.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5613C00001
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: Hyperphosphatemia
Keywords: S-phosphate, hyperphosphatemia, hemodialysis, ESRD
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 mg bid (Experimental): 1 mg AZD1722 bid
  Interventions: Drug: AZD1722
- 3 mg bid (Experimental): 3 mg AZD1722 bid
  Interventions: Drug: AZD1722
- 10 mg bid (Experimental): 10 mg AZD1722 bid
  Interventions: Drug: AZD1722
- 30 mg bid (Experimental): 30 mg AZD1722 bid
  Interventions: Drug: AZD1722
- 3 mg od (Experimental): 3 mg AZD1722 od
  Interventions: Drug: AZD1722
- 30 mg od (Experimental): 30 mg AZD1722 od
  Interventions: Drug: AZD1722
- Placebo (Placebo Comparator): Placebo (double dummy technique)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1722 — AZD1722, oral tablet
  Arms: 1 mg bid; 10 mg bid; 3 mg bid; 3 mg od; 30 mg bid; 30 mg od
Drug: Placebo — Placebo bid, double dummy technique
  Arms: Placebo

SUMMARY:
Randomized. double blind, placebo controlled, parallel arms dose finding study with a 4 weeks treatment period

DETAILED DESCRIPTION:
The study consists of a screening period of approximately 1 week, a wash out period of up to 3 weeks, where existing phosphate lowering medication is withheld, a 4-week treatment period and a follow-up period of up to 2 weeks, during which patients are put back on their pre washout phosphate lowering medication.

The wash out period will be either 1 week, 2 weeks or 3 weeks depending on the increase in s-phosphate levels.

There are 7 parallel treatment arms in the study with bid and od treatment regimens.

Laboratory efficacy endpoints and safety assessments will be evaluated at various times throughout the study.

The target population of the study is: male or female patients, above18 years of age with End Stage Renal Disease (ESRD) on chronic maintenance hemodialysis (HD) 3 times a week for a minimum of 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males aged ≥18 years
2. Chronic maintenance hemodialysis 3 x/week for a at least 3 months
3. Prescribed and taking at least 3 doses of phosphate binder per day
4. Serum phosphate levels should be between 3.5 and 8.0 mg/dL ; 1.13 mmol/L and 2.58 mmol/L (inclusive) at screening
5. Total serum calcium levels 2.0 - 2.6 mmol/L inclusive at screening
6. For randomization in the study, after up to 3 weeks wash out of phosphate binders, patients must have serum phosphate levels of at least 6. 0 mg/dL (1.94 mmol/L) but below 10 mg/dL (3.23 mmol/L) and have had an increase of at least 1.5 mg/dL (0.48 mmol/L) vs pre wash out

Exclusion Criteria:

1. Severe hyperphosphatemia defined as >10 mg/dL on Phosphate-binders at all time points during clinical routine monitoring for the 3 preceding months before screening visit.
2. Serum parathyroid hormone >1200 pg/mL
3. Significant metabolic acidosis
4. Clinical signs of hypovolemia at randomization

   -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrology PC, Denver, CO 80230
Locations (41):
- United States (16):
  - Research Site, Downey, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Flushing, New York
  - Research Site, Maspeth, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, San Antonio, Texas
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Częstochowa
  - Research Site, Działdowo
  - Research Site, Legnica
  - Research Site, Lublin
  - Research Site, Radom
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zamość
  - Research Site, Zgierz
  - Research Site, Żary
- Slovakia (7):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Hlohovec
  - Research Site, Košice
  - Research Site, Piešťany
  - Research Site, Púchov
  - Research Site, Senica
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Doncaster
  - Research Site, Exeter
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, London

REFERENCES:
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Block GA, Rosenbaum DP, Yan A, Greasley PJ, Chertow GM, Wolf M. The effects of tenapanor on serum fibroblast growth factor 23 in patients receiving hemodialysis with hyperphosphatemia. Nephrol Dial Transplant. 2019 Feb 1;34(2):339-346. doi: 10.1093/ndt/gfy061. PMID 29617976

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg Bid: 1 mg AZD1722 bid
  AZD1722: tenapanor, oral tablet
- 3 mg Bid: 3 mg AZD1722 bid
  AZD1722: tenapanor, oral tablet
- 10 mg Bid: 10 mg AZD1722 bid
  AZD1722: tenapanor, oral tablet
- 30 mg Bid: 30 mg AZD1722 bid
  AZD1722: tenapanor, oral tablet
- 3 mg od: 3 mg AZD1722 od
  AZD1722: tenapanor, oral tablet
- 30 mg od: 30 mg AZD1722 od
  AZD1722: tenapanor, oral tablet
Period: Overall Study
Arm/Group | 1 mg Bid | 3 mg Bid | 10 mg Bid | 30 mg Bid | 3 mg od | 30 mg od | Placebo
Started | 23 | 21 | 23 | 26 | 22 | 21 | 26
Completed | 18 | 13 | 19 | 13 | 18 | 12 | 22
Not Completed | 5 | 8 | 4 | 13 | 4 | 9 | 4
Not completed — Adverse Event | 5 | 4 | 3 | 10 | 2 | 8 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg Bid | 3 mg Bid | 10 mg Bid | 30 mg Bid | 3 mg od | 30 mg od | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 23 | 26 | 22 | 21 | 26 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (14.79) | 61.5 (11.21) | 62.7 (12.53) | 59.7 (12.96) | 57.6 (15.78) | 58.2 (15.75) | 56.1 (13.14) | 59.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 15 | 17 | 12 | 13 | 16 | 104
  Male | 7 | 6 | 8 | 9 | 10 | 8 | 10 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 10 | 4 | 8 | 6 | 6 | 48
  Not Hispanic or Latino | 16 | 14 | 13 | 22 | 14 | 15 | 20 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 8
  Asian | 1 | 0 | 3 | 1 | 1 | 0 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 8 | 3 | 9 | 6 | 3 | 4 | 35
  White | 17 | 12 | 16 | 15 | 13 | 16 | 17 | 106
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 3
serum phosphorus [Mean (Standard Deviation); unit: mg/dL] | 7.55 (1.003) | 7.92 (1.005) | 7.32 (1.063) | 7.76 (1.183) | 7.73 (1.276) | 7.61 (0.847) | 7.87 (1.488) | 7.68 (1.124)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphate Levels
Description: Change in serum phosphate levels from the end of wash out (pre randomization value) to end of treatment
Time Frame: End of wash out (pre randomization value) to end of treatment (Day 29)
Population: two patients in the 30 mg bid group are not included in the analysis since they had no post randomization serum phosphorus measurements
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1 mg Bid | 3 mg Bid | 10 mg Bid | 30 mg Bid | 3 mg od | 30 mg od | Placebo
Number analyzed (Participants) | 23 | 21 | 23 | 24 | 22 | 21 | 26
mg/dL | -.47 (1.553) | -1.18 (1.391) | -1.7 (2.018) | -1.98 (2.007) | -.56 (1.763) | -1.11 (1.469) | -.54 (1.802)
Statistical Analysis 1: Comparison: 1 mg Bid vs 3 mg Bid vs 10 mg Bid vs 30 mg Bid vs 3 mg od vs 30 mg od vs Placebo; Test type: Superiority; p = 0.012, ANCOVA

2. Secondary Outcome: Change From Baseline in Calcium x Phosphorus Product
Description: Change from baseline (end of wash out) in calcium x phosphorus product
Time Frame: End of wash out (pre randomization value) to end of treatment (Day 29)
Population: The number of patients analyzed are less than the randomized number since the data to accomplish the analysis was not available.
Measure: Mean (Standard Deviation); unit: mg/dL * mg/dL
Arm/Group | 1 mg Bid | 3 mg Bid | 10 mg Bid | 30 mg Bid | 3 mg od | 30 mg od | Placebo
Number analyzed (Participants) | 22 | 19 | 20 | 23 | 21 | 20 | 24
mg/dL * mg/dL | -5.16 (9.75) | -12.02 (14.02) | -12.44 (15.94) | -16.6 (18.01) | -3.59 (18.59) | -11.02 (11.57) | -2.50 (13.67)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a total of 5 weeks; 4-weeks of treatment and 1 treatment-free week
Arm/Group | 1 mg Bid | 3 mg Bid | 10 mg Bid | 30 mg Bid | 3 mg od | 30 mg od | Placebo
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/21 | 0/23 | 0/26 | 0/22 | 0/21 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/21 | 3/23 | 2/26 | 1/22 | 0/21 | 4/26
Other Adverse Events (participants affected / at risk) | 6/23 | 6/21 | 11/23 | 17/26 | 4/22 | 11/21 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Bid (N=23) | 3 mg Bid (N=21) | 10 mg Bid (N=23) | 30 mg Bid (N=26) | 3 mg od (N=22) | 30 mg od (N=21) | Placebo (N=26)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Bid (N=23) | 3 mg Bid (N=21) | 10 mg Bid (N=23) | 30 mg Bid (N=26) | 3 mg od (N=22) | 30 mg od (N=21) | Placebo (N=26)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 11 (11) | 17 (17) | 4 (4) | 11 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days